CLINICAL TRIAL: NCT02963870
Title: Randomized Controlled Trial of the Effectiveness of the Cognitive-behavioral Approach, Standard Plan Security on Relapse Suicidal Adolescents
Brief Title: The Cognitive-behavioral Approach, Standard Plan Security on Relapse Suicidal Adolescents
Acronym: SECURIPLAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2015_843_0009
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Treatment of Suicidal Recidivism in Adolescents Population
Keywords: Cognitive behavioral; security plan; suicidal Recidivism in adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- security plan (Experimental): groups of adolescents aged 12-17 hospitalized for TS and randomized to a group treated with security plan and the usual treatment
  Interventions: Other: Security Plan
- standard treatment only. (Active Comparator): group receiving standard treatment only.
  Interventions: Other: Security Plan

INTERVENTIONS:
Other: Security Plan — This study compared two groups of adolescents aged 12-17 hospitalized for TS and randomized to a group treated with the Security Plan plus the usual treatment and a group receiving standard treatment only.

SUMMARY:
The recommendation for the treatment of suicidal adolescents, Cognitive Behavioral Therapy (CBT) targeted new generation offer effective approaches to suicidal crisis and relapse prevention

DETAILED DESCRIPTION:
The recommendation for the treatment of suicidal adolescents, Cognitive Behavioral Therapy (CBT) targeted new generation offer effective approaches to suicidal crisis and relapse prevention.

Since 2009, our team is engaged in a partnership between France and Quebec Interuniversity agreement concluded by a University Picardie Jules Verne-University of Montreal. In this context, two teams G4 (Amiens and Rouen) have received training in suicidal crisis, including the security plan by a university instructor and TCC Québec, Dr. Labelle. Furthermore, we complete a descriptive and prospective study of risk and protective factors for adolescent suicide in which the Quebec team of Professor Labelle contributes as an expert (sponsor: Rouen). 200 subjects were recruited on 2 years by 3 (CHU Amiens, CH Compiègne, CHU Rouen) with an assessment of recurrence at 1 year (lost rates of view = 15%). The first results highlight the central role of personal coping strategies (coping) in suicidal recurrence. We want extend this study to validate the implementation of the security plan (safety level) with suicidal adolescents. The security plan is the initial step of the TCC approach short of suicidal crisis. It is established after working with adolescents and their families (chain analysis of the suicidal crisis, coping self-evaluation and identification of support resources). Developed by Stanley B from Columbia University and adapted for francophone adolescents R Labelle and JJ Breton wrote this list those resources and coping strategies to apply in case ideation and suicidal crisis. Signed by the young person and his family, he then uses to frame the monitoring and management plan of the youth and his family environment, friendly and professional in case of suicidal crisis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 12 and 17, boys and girls, hospitalized for attempted suicide
* Adolescents whose parents gave informed consent and who themselves expressed their willingness to participate in research.
* Patients covered by the social insurance system

Exclusion Criteria:

* Clinical situations with self-injury without suicidal intent or suicide attempt
* mental disorders significantly impair the self-assessment questionnaire capacities: Intellectual disability, autism spectrum disorder, acute psychotic state and, psychopathy (including assessment questionnaire Frick) and the active use of alcohol and toxic (DEP teen> 20)
* have benefited a security plan before the study
* adolescents deprived of liberty.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of suicide attempt | 12 months
  Occurrence of suicide attempt recurrence (documented by CNRS) during the year following randomization.

SECONDARY OUTCOMES:
Occurrence of relapse Suicide attempt | 6 months
  Occurrence of relapse Suicide attempt within 6 months of randomization.
Observance | 6 months and 12 months
  Observance at 6 months and 1 year using the categories used in the Giraud study
coping strategies of the adolescent | 12 months
  Compare at 1 year the evolution of coping strategies of the adolescent assessed by changes in coping scores assessed by self-questionnaire Friedenberg (ACS) from randomization to 1 year later.
Evolution of social support perceived by the teen evaluat | 12 months
  Compare at 1 year evolution of social support perceived by the teen evaluated by varying the scores of self-questionnaire Sarason (SSQ6) from randomization to 1 year later.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc GUILE, professor, Study Director — CHU amiens-Picardie; LEGRAND, Doctor, Principal Investigator — CHP Philippe Pinel Amiens; GERARDIN, Doctor, Principal Investigator — University Hospital, Rouen; BALEYTE, Doctor, Principal Investigator — University Hospital, Caen; Bernadette BAKHACHE, Doctor, Principal Investigator — CH St-Quentin; Maud PERCQ, Doctor, Principal Investigator — EPSMD Aisne; VERVEL, Doctor, Principal Investigator — CH Compiègne
Locations (3):
- France (3):
  - Chu Amiens Picardie, Amiens
  - CHU CAEN, Caen
  - Chu Charles Nicolle, Rouen